CLINICAL TRIAL: NCT01925378
Title: A PHASE II SINGLE-ARM INTERVENTION TRIAL OF NELFINAVIR IN PATIENTS WITH GRADE 2/3 or 3 CERVICAL INTRAEPITHELIAL NEOPLASIA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is going to open in a new site
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Joseph Anthony Lucci III, Professor and Director Division of Gynecologic Oncology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110917-01
Record Dates: First submitted 2013-04-30; First posted 2013-08-19 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Cervical Dysplasia
Keywords: Cervical Dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nelfinavir (Experimental): This is a single arm intervention trial of nelfinavir in women with grade 2/3 or grade 3 cervical intraepithelial neoplasia
  Interventions: Drug: Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir — All medications which a patient is taking will be reviewed at each visit, including the screening, day 1, weeks 4,12, 24.
  All patients enrolled in the study will receive 1,250 mg twice PO daily for a 24 week duration.
  Other Names: Viracept

SUMMARY:
Preliminary data showed that Nelfinavir has selective apoptotic effects on HPV+ cervical tumor cell lines. Furthermore, in a Phase I clinical trial, the combination of NFV and chemoradiotherapy showed acceptable toxicity and promising activity in patients with pancreatic cancer. Therefore, for the proposed research, the principal investigator will use a single-arm Phase II intervention trial study design with focus on the efficacy of NFV to induce complete or partial remission of CIN 2/3 or CIN 3 as well as biomarker evaluation.

DETAILED DESCRIPTION:
2.0 BACKGROUND AND RATIONALE 2.1 Cervical Cancer Etiology and Targets for Intervention Cervical cancer is one of the most common causes of cancer-related deaths in women worldwide. Implementation of widespread screening has created drastic improvements in the incidence of cervical cancer as well as significant decreases in mortality over the last 30 years. It is estimated that in 2011, there will be 12,710 women in the US diagnosed with cervical cancer and ultimately 4,290 women will die from the disease. Cervical cancer is unique in that there exists a well-defined pre-malignant phase, referred to as cervical dysplasia, which can be suspected on cytological examination (pap smear) of exfoliated cervical cells and confirmed on histological examination of cervical biopsy material. The pre-cancerous changes represent a spectrum of histological abnormalities or cervical intraepithelial neoplasia (CIN) ranging from CIN 1 (mild dysplasia) to CIN2 (moderate dysplasia) to CIN3 (severe dysplasia/ carcinoma in situ). The timeline of progression for CIN 3 to invasive cancer in untreated women averages between 8.1 and 12.6 years.The surgical treatment of cervical pre-cancerous is therapeutically efficacious. However, it is an invasive procedure which has been associated with fertility and obstetrical complications in reproductive aged women. An attractive alternative to an excisional or ablative procedure would be to utilize an agent which could be applied topically or taken by mouth to foster regression of cervical dysplasia. The use of natural, synthetic, or biologic chemical agents to reverse, suppress, or prevent carcinogenic progression is called chemoprevention.

A prerequisite for cervical cancer is persistent infection by a high-risk human papillomavirus allowing viral gene products sufficient time with which to induce carcinogenesis through a generally well understood natural history. Cancer-associated HPV types encode three oncogenes, E5, E6 and E7, and the E6 and E7 proteins have a significant role in malignant transformation. E6 and E7 stimulate cell proliferation by interfering with the function of regulatory proteins in cells, including the tumor suppressors p53 and pRB. Co-expression of both E6 and E7 leads to indefinite proliferation and immortalization of keratinocytes and induces premalignant neoplasms. HPV-E5, a transmembrane protein, can activate PI3K-Akt signalling. The up-regulation of PI3K-Akt survival signaling protects HPV-16 E5-expressing cells from apoptosis induced by ultraviolet irradiation. The major transforming capability of HPV is dependent on E6 and E7. However, E5 is necessary for full activation of E7, and the induction of PI3K-Akt-dependent apoptotic inhibition by E5 contributes to E7-mediated oncogenesis.

The work done to evaluate PI3K activity as a potential marker of CIN progression further supports the idea that this pathway is also up-regulated in pre-cancerous lesions. The catalytic subunit alpha of PI3K is expressed in non-invasive cervical lesions and has shown potential as a carcinogenesis-related marker for early intraepithelial lesion of the uterine cervix in cytology samples. Among other potential markers, PIK3CA showed a superior specificity to distinguish CIN3 from other groups. Yao et al 2008 showed that positive rates of PI3K and Akt were significantly lower in normal cervical epithelium and cervical intraepithelial neoplasia than in cervical carcinoma (0.0% and 42.9% vs. 69.7%, P<0.01; 10.0% and 52.4% vs. 75.0%,P<0.01). Specifically, PI3K/Akt activation increased with grade of dysplasia with invasive carcinoma having the highest activity. They also showed that expression of PI3K protein positively correlated to the expression of Akt protein(r=0.425, P<0.01).

2.2 Nelfinavir (NFV) Background Nelfinavir (NFV) induces cell cycle arrest, endoplasmic reticulum stress, autophagy, and apoptosis is cancer cells. As a protease inhibitor used in patients with HIV, NFV predominately targets proteases 1 and 2, but it is also known that part of the efficacy is due to selective inhibition of the proteosome. The pathogenecity of high risk HPV is dependent on expression of viral E6 proteins which inappropriately activate the 26S proteosome to degrade p53 and other cellular proteins that are detrimental to viral replication; specific HIV protease inhibitors can block the ability of HPV16 E6 to degrade p53 and selectively kill E6-dependent cervical carcinoma cells. Furthermore, HIV protease inhibitors have been shown to inhibit the PI3K/Akt signaling pathway with NFV being the most potent. NFV's mechanism of action involves decreasing Akt phosphorylation. In addition, at concentrations (micromolar) achievable in the serum of patients taking usual dosing of the drug (1250mg PO BID), Akt phosphorylation is inhibited. At our institution, we have shown that HPV-infected cervical cancer cells lines treated with NFV underwent apoptosis and decreased cell proliferation in a dose dependent manner. Furthermore, we have shown through a recent retrospective study that HIV-infected women with cervical dysplasia who were treated with protease inhibitors (PI), including NFV were more likely to regress than those not on a PI-containing regimen.

Because PI3K/Akt is up-regulated in CIN2/3 and NFV has been shown to inhibit this pathway in HPV-infected cervical cancer cell lines, we aim to further evaluate the effectiveness of NFV as an intervention for CIN2/3 and correlate these findings with phospho-Akt levels in cervical tissue. Several intervention trials have been conducted in women with CIN using retinoids, ß-carotene, difluoromethylornithine, and indole-3- carbinol and over 300 women with CIN 3 were followed in these trials for one to 15 months while none of them developed invasive cervical cancer. Therefore, this proposed intervention trial of 24 weeks (6 months) duration should allow a safe evaluation of NFV as a potential agent for a future randomized Phase III trial.

Development of a new drug for cancer treatment is expensive and time consuming. Repositioning of a drug which is already FDA approved for another indication allows for more rapid evaluation and potential implementation of a novel cancer therapy. NFV has been identified to have anti-cancer effects in vitro, and compared to other protease inhibitors it is more potent in causing cell death. NFV has over 10 years of safety and pharmacokinetic data in HIV-infected individuals. Standard dosing for the treatment of HIV is 1,250 mg PO BID, and this dose has demonstrated plasma concentrations in vivo which correlate with necessary concentrations of successful in vitro studies. Furthermore, evaluation of the standard dose offers the availability of commercially produced tablets, the known and acceptable side effect profile, and the ease of twice daily dosing. For these reasons NFV is an excellent candidate for repositioning as an intervention for cervical dysplasia, which can be quickly evaluated in this phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Cytology report with a High Grade Squamous Intra Epithelial Lesion "HSIL" or have histologically proven CIN 2/3 or CIN 3 diagnosed by cervical biopsy between 2 and 8 weeks prior to enrollment. For a patient to be eligible, the Cytology report must state High Grade Squamous Intra Epithelial Lesion "HSIL" or the pathology report must clearly state "CIN 2/3" or "CIN 3" or must state "moderate-severe dysplasia", "moderate severe dyskaryosis," "severe dysplasia," or "severe dyskaryosis." Patients with a diagnosis of CIN 2 alone or moderate dysplasia or dyskaryosis alone are not eligible for this study.
* Patients must be at least 18 years of age.
* Patients must have a satisfactory (readable, good quality) colposcopic evaluation at least 14 days after diagnostic biopsy.
* Patients must have colposcopically visible cervical lesion at entry consistent with biopsy.
* Patients must have a negative urine pregnancy test within 14 days of starting the NFV. Women of childbearing potential must practice an acceptable form of contraception (e.g. intrauterine device, contraceptive pills, diaphragm, condoms).
* Patients must have a GOG Performance Status of 0, 1, or 2.
* Patients must be good candidates for delayed treatment of their CIN, i.e. they must be reliable to return for follow-up and provide a combination of at least three phone numbers or addresses for contact.
* Patients must have adequate*:
* CBC/Platelets: Hemoglobin (HgB) greater than 10.0g/dl; white blood cell (WBC) count greater than 3000/mcl; Platelet count greater than 125,000/mcl.
* Renal function: Creatinine less than or equal to 1.5 x Upper Limit Normal (ULN).
* Hepatic function: Total bilirubin less than or equal to 1.5 x ULN excluding Gilbert's disease; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.0 x ULN.
* Glycemic control: fasting glucose < 126; random glucose <200; hemoglobin A1C ≤ 7.0%

  *These lab results must be evaluated prior to patient enrollment.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.
* Patients must have a negative HIV test within 14 days of starting the NFV.
* Patients with allergies or known sensitivity to Nelfinavir will be excluded or withdrawn after treatment, if deemed a safety concern by the principal Investigator.

Exclusion Criteria:

Ineligible Patients

* Patients who are pregnant or breast-feeding.
* Patients with cytologic or biopsy evidence of endocervical dysplasia or invasive cancer.
* Patients with undiagnosed abnormal vaginal bleeding.
* Patients with a known immunocompromised condition or a positive HIV test. Patients with a prior history of cervical cancer.
* Patients with a chronic or acute renal, or hepatic disorder, a significant bleeding disorder, or any other condition which in the Investigator's opinion might preclude study participation for the duration of the trial.
* Patients taking concurrent medication that is metabolized by the CYP3A4 isoenzyme.
* Patients taking the following concurrent medications: astemizole, cisapride, salmeterol, alfuzosin, terfinadine, amiodarone, midazolam, quinadine, ergot derivatives, pimozide, rifampin, triazolam, warfarin, azithromycin, carbamezpine, cyclosporine, didanosine, fluticasone propionate, phenobarbital, phenytoin, trazadone, sirolimus, tacrolimus , and St. John's wart.
* Patients who are unwilling, or unable, to practice an acceptable form of contraception (e.g. intrauterine device, contraceptive pills, diaphragm, condoms). For those women who choose to use oral contraceptive pills, they will be encouraged to use a second form of contraception, such as condoms, because of the potential for altered serum levels of oral contraceptives.
* Patients with uncontrolled diabetes; as defined by hemoglobin A1C ≥ 7.1%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
1.1 Efficacy of Nelfinavir (NFV) to induce complete remission (or partial regression to CIN 1) of CIN 2/3 or CIN 3 as evaluated in the post-treatment excisional biopsy. | 24 weeks
  EVALUATION CRITERIA
  Parameters of response:
  Histologic evaluation of the post-treatment LLETZ/cone specimen.
  (1) Persistent with worst disease being CIN 3; (2) Persistent with worst disease being CIN 2/3; (3) Persistent with worst disease being CIN 2; (4) Persistent with worst disease being CIN 1; (5) Normal tissue; no evidence of CIN present; (6) Squamous cell carcinoma, in situ.
  Histologic Complete Response will be judged as complete absence of any histologic evidence of CIN in the biopsy or LLETZ .
  Histologic Partial Response will be judged as regression of CIN 2/3 or CIN 3 to persistent disease with worst grade being CIN 1 in the LLETZ cone biopsy.
  Histologic Persistent Disease will be defined as evidence of CIN 2, CIN 2/3 or CIN 3 in the LLETZ/cone biopsy.
  Histologic Progression: Evidence of disease progression such as invasive carcinoma.

SECONDARY OUTCOMES:
targeted mechanism of NFV in histological response | 24 weeks
  Pathway inhibition will be demonstrated when there is a decrease of PI3K and/or Akt on IHC between the enrollment biopsy and the final biopsy or the LLETZ/cone specimen

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Lucci, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] Hampson L, Kitchener HC, Hampson IN. Specific HIV protease inhibitors inhibit the ability of HPV16 E6 to degrade p53 and selectively kill E6-dependent cervical carcinoma cells in vitro. Antivir Ther. 2006;11(6):813-25. PMID 17310826
- [Background] Pisani P, Bray F, Parkin DM. Estimates of the world-wide prevalence of cancer for 25 sites in the adult population. Int J Cancer. 2002 Jan 1;97(1):72-81. doi: 10.1002/ijc.1571. PMID 11774246
- [Background] Siegel R, Ward E, Brawley O, Jemal A. Cancer statistics, 2011: the impact of eliminating socioeconomic and racial disparities on premature cancer deaths. CA Cancer J Clin. 2011 Jul-Aug;61(4):212-36. doi: 10.3322/caac.20121. Epub 2011 Jun 17. PMID 21685461
- [Background] Solomon D, Schiffman M, Tarone R; ALTS Study group. Comparison of three management strategies for patients with atypical squamous cells of undetermined significance: baseline results from a randomized trial. J Natl Cancer Inst. 2001 Feb 21;93(4):293-9. doi: 10.1093/jnci/93.4.293. PMID 11181776
- [Background] Sporn MB. Approaches to prevention of epithelial cancer during the preneoplastic period. Cancer Res. 1976 Jul;36(7 PT 2):2699-702. PMID 1277177
- [Background] Walboomers JM, Jacobs MV, Manos MM, Bosch FX, Kummer JA, Shah KV, Snijders PJ, Peto J, Meijer CJ, Munoz N. Human papillomavirus is a necessary cause of invasive cervical cancer worldwide. J Pathol. 1999 Sep;189(1):12-9. doi: 10.1002/(SICI)1096-9896(199909)189:13.0.CO;2-F. PMID 10451482
- [Background] Zhang L, Epstein JB, Poh CF, Berean K, Lam WL, Zhang X, Rosin MP. Comparison of HPV infection, p53 mutation and allelic losses in post-transplant and non-posttransplant oral squamous cell carcinomas. J Oral Pathol Med. 2002 Mar;31(3):134-41. doi: 10.1034/j.1600-0714.2002.310302.x. PMID 11903818